CLINICAL TRIAL: NCT05507502
Title: Optimizing the Timing of Influenza Vaccination in Patients With Heart Failure: the FLU-HF Randomized Trial: a Randomized Controlled Trial
Brief Title: Timing of Influenza Vaccination in Patients With Heart Failure
Acronym: FLU-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abhinav Sharma (Other)
Responsible Party: Sponsor-Investigator, Abhinav Sharma, Assistant Professor, Division of Cardiology, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-7425
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 manner to receiving the influenza vaccination during their heart failure hospitalization versus receiving the vaccine during their first follow-up in the heart failure clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-patient vaccination arm (Active Comparator): Participants in this arm will receive the influenza vaccination during their heart failure hospitalization.
  Interventions: Biological: Influenza vaccination administration
- In-clinic vaccination arm (Active Comparator): Participants in this arm will receive the influenza vaccination during their follow up visit in the heart failure clinic 30 days post-discharge.
  Interventions: Biological: Influenza vaccination administration

INTERVENTIONS:
Biological: Influenza vaccination administration — There will be approximately 40 participants who consent; they will be randomized in a 1:1 manner to receiving the influenza vaccination during their heart failure hospitalization versus receiving the vaccine during their first follow-up in the heart failure clinic.

SUMMARY:
Heart failure (HF) is one of the most common causes of hospital admission in Canada and costs the Canadian healthcare system over $1 billion annually. Influenza vaccination is an inexpensive strategy to prevent influenza infections and reduce an important trigger for HF decompensation and hospital readmission. Yet, the optimal timing of vaccine administration remains unclear. When patients with HF are admitted to the hospital with an acute decompensation in advance of, or during, the 'flu season', this can be an ideal time to administer the vaccine. However, patients with acute HF decompensation have significant inflammatory injury, and may have substantially impaired immune responses; thus vaccine administration while admitted during an acute decompensated HF episode may not lead to high anti-influenza antibody titres. A more effective strategy can be to vaccinate after the decompensation has resolved, when patients are more stable. The FLU-HF randomized trial will determine whether administering the influenza vaccine to patients admitted in-hospital with an acute HF decompensation or waiting until they have stabilized as an out-patient leads to an improved anti-influenza response.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Admitted in hospital with primary diagnosis of acute HF
* Prior diagnosis of chronic HF > 3 months prior to admission
* Not on inotropes, mechanical support, or IV diuretics for 24 hours
* Able to follow-up within the MUHC HF clinic as per schedule
* agree to receive influenza vaccination

Exclusion Criteria:

* Any person who does not meet the above criteria and/or who refuses to participate
* Already received this seasons influenza vaccination
* Known allergy to influenza vaccination or components of the influenza vaccination
* Unlikely to survive to discharge as per admitting physician
* Prior organ transplant
* Undergoing chemotherapy for active malignancy
* Currently randomized in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion for one or more strains in the influenza vaccine one month following vaccination. | Randomization to one month post randomization
  Seroconversion will be measured by antibody as assessed by the hemagglutination inhibition (HI) assay.

SECONDARY OUTCOMES:
Change in NTproBNP | Randomization to one month post randomization
  Serologic blood work measured at randomization and post-randomization
Change in high-sensitivity troponin | Randomization to one month post randomization
  Serologic blood work measured at randomization and post-randomization
Changes in inflammatory markers | Randomization to one month post randomization
  Inflammatory markers as measured by HsCRP, IL1, IL6, at randomization and post-randomization

OTHER OUTCOMES:
Seroconversion for one or more strains in the influenza vaccine upto three months following vaccination. | Randomization to three months post randomization
  Seroconversion will be measured by antibody as assessed by the hemagglutination inhibition (HI) assay.
Change in NTproBNP | Randomization to three months post randomization
  Serologic blood work measured at randomization and post-randomization
Change in high-sensitivity troponin | Randomization to three months post randomization
  Serologic blood work measured at randomization and post-randomization
Changes in inflammatory markers | Randomization to three months post randomization
  Inflammatory markers as measured by HsCRP, IL1, IL6, at randomization and post-randomization

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided